CLINICAL TRIAL: NCT06136910
Title: Oncorine (H101) Combined With Tislelizumab and Platinum-based Two-drug Chemotherapy in Previously Untreated Advanced Non-small Cell Lung Cancer, a Phase II Single-arm Clinical Trail
Brief Title: Oncorine (H101) Combined With Tislelizumab and Chemotherapy in Previously Untreated Advanced Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCOG006
Record Dates: First submitted 2023-11-07; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Untreated Advanced Non-small Cell Lung Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- H101 combined with tirilizumab and platinum-containing two-drug chemotherapy (Experimental): 1. Recombinant human adenovirus type 5 injection(H101), intratumoural, administered for 4 cycles, 1 injection on day 1 (d1) of each cycle.The number of injections should be determined according to the patient's tolerance and the ease of manipulation of the injection site, and should be no less than 2 times.
  2. Tirilizumab injection, 200 mg, IV, d1, Q21d, administered until disease progression or intolerable side effects occur
  3. Platinum-containing two-agent chemotherapy Adenocarcinoma: pemetrexed plus carboplatin Non-adenocarcinoma: paclitaxel/gemcitabine combined with carboplatin
  Interventions: Drug: Recombinant human adenovirus type 5 injection (H101) combined with tirilizumab and platinum-containing two-drug chemotherapy

INTERVENTIONS:
Drug: Recombinant human adenovirus type 5 injection (H101) combined with tirilizumab and platinum-containing two-drug chemotherapy — 1. Recombinant human adenovirus type 5 injection : 21 days is one treatment cycle, in principle, 4 cycles of administration, 1 injection on day 1 (d1) of each cycle; the number of injections is determined according to the patient's tolerance and the ease of operation of the injection site, no less than 2 times.
  2. tirelizumab: 200mg intravenous, d1, Q21d, administered until disease progression or intolerable side effects occur
  3. platinum-containing two-drug chemotherapy: adenocarcinoma, pemetrexed combined with carboplatin, 4-6 cycles, d2, Q21d; non-adenocarcinoma, paclitaxel/gemcitabine combined with carboplatin, 4-6 cycles, d2, Q21d.

SUMMARY:
This is a single-arm, single-centre phase II study to evaluate the efficacy (PFS, ORR, DCR) and safety of recombinant human adenovirus type 5 in combination with tirelizumab and platinum-containing dual-agent chemotherapy in previously untreated patients with advanced non-small cell lung cancer who are EGFR/ALK negative. The study is divided into 2 phases.

DETAILED DESCRIPTION:
Phase 1 is a preliminary exploration of safety and efficacy. The safety and efficacy of the regimen was assessed in the 10 patients enrolled for interim analysis. Phase 2 will continue to expand the sample size to assess the efficacy and safety of the regimen, with 20 patients planned to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Fully informed about the study and voluntarily signed an informed consent form (ICF); ≥18 years and ≤75 years;
2. ECOG score 0-1;
3. non-small cell lung cancer (NSCLC) confirmed by histology or pathology;
4. stage IV on imaging assessment;
5. no EGFR or ALK gene mutations (genetic testing may not be performed in patients with squamous lung cancer);
6. no previous antitumour treatment for NSCLC No prior antitumour therapy for NSCLC;
7. lesions suitable for intratumour injection of drugs;
8. measurable or assessable lesions according to RECIST 1.1 criteria.

Exclusion Criteria:

1. histological or cytological pathology of the tumour confirms a combined small cell lung cancer component;
2. those with tests suggesting severe organ dysfunction;
3. subjects with any active, known or suspected autoimmune disease are excluded;
4. expected survival is less than 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2024-05-09 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The time from the date of first treatment to the first occurrence of disease progression or death from any cause, whichever event occurs first. | 1 year
  Progression-free survival (PFS) as assessed by the investigators according to RECIST 1.1 criteria

SECONDARY OUTCOMES:
Proportion of CR and PR in all patients. | 1 year
  Objective response rate: ORR
Proportion of CR, PR and SD in all patients. | 1 year
  Disease control rate: DCR
Safety statistics will be analysed for adverse events. | 1 year
  Safety statistics will be analysed for adverse events, including AEs, SAEs, drug-related AEs, AEs leading to dose adjustments, and AEs leading to withdrawal from the trial.All adverse events will also be rated based on the NCI CTCAE version 5.0, and AEs greater than or equal to grade 3 will be statistically summarised.

CONTACTS AND LOCATIONS:
Overall Officials: Liyun Miao, Doctor, Study Chair — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School; Dongyong Yang, Bachelor, Study Chair — The Second Attached Hospital Of Fujian Medical University; Jianhong Xiao, Bachelor, Study Chair — MinDong Hospital of Ningde City; Minlin zheng, Bachelor, Study Chair — The Second Hospital of Zhangzhou
Locations (1):
- Fujian Cancer Hospital, Fuzhou, Fujian, China